CLINICAL TRIAL: NCT00683072
Title: Patient-Ventilator Dyssynchrony: How is the Effect of Management?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Other Study IDs: NCKUH-9703023
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Respiratory Failure
Keywords: Ventilator; patient-ventilator asynchrony
MeSH Terms: conditions — Respiratory Insufficiency; Patient-Ventilator Asynchrony

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1

SUMMARY:
Although patient-ventilator asynchrony is a frequent phenomenon, its course following management is unknown. As the aid of a data recording system, we try to observe the consequence of patient-ventilator asynchrony following management. Our target is aimed at the patients with high asynchronization index ( > 10%) as this group of patients have been shown to have prolonged course in intensive care unit and are also prone to be tracheostomized

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to respiratory intensive care unit with acute respiratory failure and presence of patient-ventilator asynchrony(AI of more than 10%)
* patient can trigger the ventilator

Exclusion Criteria:

* High oxygen fraction: > 60%.
* High PEEP need: > 12cmH2O.
* Hemodynamic unstable: shock
* Central nervous system problem.
* Hyperacitve delirium
* Without informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between March 2008 through December 2008, patients admitted to our respiratory intensive care unit for the management of acute respiratory failure were daily screened for the presence of patient-ventilator asynchrony.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Asynchrony index (AI). (Number of asynchrony events/total respiratory rate) | 20 minutes after alternation of ventilator settings or any therapeutic means

CONTACTS AND LOCATIONS:
Overall Officials: Chang wen Chen, MD, MS, Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan